CLINICAL TRIAL: NCT03550677
Title: Effect of Intraoperative Ankle Nerve Blocks on Postoperative Discharge in Patients Undergoing Orthopaedic Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Ceyda Ozhan Caparlar, Anesthesiology Specialist, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 49/07
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Operative Incision
Keywords: Ankle nerve block; post operative analgesia; patient satisfaction; foot surgery
MeSH Terms: conditions — Surgical Wound; Patient Satisfaction | interventions — Anesthesia, General; Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group General Anesthesia (Experimental): These group patients will be monitored with ECG, pulse oximetry and noninvasive blood pressure. Anesthesia will be induced using 2-2.5 mg/kg propofol, 1-2 mcg/kg fentanyl, 10 mg-20 mg rocuronium and a proper size laryngeal mask airway will be placed to secure the airway. The lungs will be ventilated with a mixture of 50% and 50% oxygen.
  Interventions: Procedure: general anesthesia
- Group Ankle Block (Experimental): These group patients will be monitored with ECG, pulse oximetry and noninvasive blood pressure. Anesthesia will be induced using 2-2.5 mg/kg propofol, 1-2 mcg/kg fentanyl, 10 mg-20 mg rocuronium and a proper size laryngeal mask airway will be placed to secure the airway. The lungs will be ventilated with a mixture of 50% and 50% oxygen. After than an ankle block will be performed in patient group block patients using a mixture of 5 ml of 2% lidocaine and 10 ml of 0.5 bupivacaine the same amount placebo (saline) in group placebo under the guidance of peripheral nerve stimulator then the anesthesia will be disconnected and LMA will be removed. The patients will be transferred from postoperative care unit toward after they are eligible for discharge according to the modified scoring system.
  Interventions: Procedure: general anesthesia; Procedure: ankle block

INTERVENTIONS:
Procedure: general anesthesia — The patient will be monitored with ECG, pulse oximetry and noninvasive blood pressure. Anesthesia will be induced using 2-2.5 mg/kg propofol, 1-2 mcg/kg fentanyl, 10-20 mg rocuronium and proper size Laryngeal mask airway will be placed securely the airway.
  Other Names: Laryngeal mask airway
Procedure: ankle block — ankle nerve block will be performed in group ankle block patients using a mixture of 5 ml of 2% lidocaine and 10 ml of 0.5% bupivacaine and same amount placebo (saline) in groups placebo under the guidance of peripheral nerve stimulator the anesthesia will be discontinued and LMA will be removed. The patients will be transferred from postoperative care unit to the ward after they are eligible for discharge according to modified Aldrete scoring system.
  Arms: Group Ankle Block

SUMMARY:
Postoperative pain is an important clinical issue which negatively affects patient's satisfaction, delays discharge and repeated admission after discharge in orthopedic surgery. Peripheral nerve blocks are commonly used for postoperative analgesia as an adjunct to analgesic drugs. The aim of this study is to evaluate the effect of ankle blocks performed at the end of the surgery on postoperative discharge times, postoperativeanalgesia, patient's satisfaction, additional analgesic requirements, and complications in patients undergoing orthopedic foot surgery.

DETAILED DESCRIPTION:
After written informed consent obtained from patients, patients will be randomly assigned to placebo group (Group I) and block group (group II) using sealed envelope method. IV venous catheter will be inserted and saline or Ringer's Lactate solution will be infused to patients for prehydration.0.1-0.5 mg/kg midazolam will be given for premedication. After arriving into OR, the patients will be monitored with ECG, pulse oximetry and noninvasive blood pressure. Anesthesia will be induced using 2-2,5 mg/kg propofol, 1-2 mcg/kg fentanyl, 10 mg-20 mg rocuronium, and a proper size laryngeal mask airway (LMA) will be placed to secure the airway. The lungs will be ventilated with a mixture of 50% air + 50% oxygen. Propofol and remifentanil based total intravenous anesthesia (TIVA) technique will be used for the maintenance of anesthesia. Tenoxicam 20 mg will be used for preemptive analgesia, cefazolin 25 mg/kg for antibiotic prophylaxis, ranitidine 50 mg for gastric protection, and metoclopramide 10 mg for postoperative nausea and vomiting. Acetaminophen 10-15 mg/kg IV will be given for postoperative analgesia at the time of wound closure.

At the end of the operation, an ankle nerve block will be performed in group II patient using a mixture of 2%lidocaine and 10 ml of bupivacaine and the same amount placebo in group I (placebo group) under the guidance of peripheral nerve stimulator. The anesthesia will be discontinued and LMA will be removed. The patients will be transferred from postoperative care unit to the ward after they were eligible for discharge according to modified Aldrete scoring system.

Postoperative analgesia will be evaluated by a study member who is blinded to study groups using visual analog scale (VAS). Acetaminophen 1000 mg p.o. were given at 8 hours intervals and an intravenous patient-controlled analgesia containing 3 mg/ml of tramadol will be used for postoperative pain therapy. Pethidine 0.5 mg/kg IV will be used for rescue analgesic if VAS score is greater than 3.

The motor block will be evaluated using Bromage scale, sensorial block with pin-prick test. The duration of motor and sensorial block, postoperative VAS scores, the time to the first analgesic requirement, total analgesic consumption and vital parameters will be recorded. Patient's satisfaction will be evaluated using 3 point scale between the scores 0 and 2. 0= poor 1= fair 2=satisfied Postoperative discharge times will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient's acceptance,
* American Society of Anesthesiologists physical status I-III
* elective orthopedic foot surgery
* general anesthesia

Exclusion Criteria:

* Pregnancy
* history of chronic pain therapy
* hypersensitivity to study drugs
* allergy to study drugs
* blood coagulation disorder
* anticoagulant use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 3 months
  Postoperative pain is evaluated using Visual Analogue Scale.

SECONDARY OUTCOMES:
postoperative discharge times | 3 months
  postoperative discharge times of paitnets after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Ozhan Caparlar, Study Director — University of Health Dıskapı Yıldırım Beyazıt Training and Hospital
Locations (1):
- University of Health Dıskapı Yıldırım Beyazıt Training and Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McLeod DH, Wong DH, Vaghadia H, Claridge RJ, Merrick PM. Lateral popliteal sciatic nerve block compared with ankle block for analgesia following foot surgery. Can J Anaesth. 1995 Sep;42(9):765-9. doi: 10.1007/BF03011173. PMID 7497554
- [Background] Fraser TW, Doty JF. Peripheral Nerve Blocks in Foot and Ankle Surgery. Orthop Clin North Am. 2017 Oct;48(4):507-515. doi: 10.1016/j.ocl.2017.06.008. Epub 2017 Aug 16. PMID 28870310